CLINICAL TRIAL: NCT04838509
Title: Diagnoses Associated With Persistent Elevation of Creatine Kinase
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Lev VOLKOV, Dr, Central Hospital, Nancy, France
Other Study IDs: 2021PI034
Record Dates: First submitted 2021-04-04; First posted 2021-04-09 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Creatine Kinase; Muscular Diseases
Keywords: Creatine Kinase
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with elevated creatine kinase
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — retrospective descriptive without intervention

SUMMARY:
Serum creatinine kinase (CK) level varies with age, gender, race and physical activity. For these reasons there is no normal serum CK level. Many pathological situations cause hyperCKemia, such as neuromuscular disorders (muscular dystrophy, inflammatory myositis, mitochondrial myopathy) and multiple systemic causes. The diagnostic approach to pauci or asymtomatic hyperCKemia can therefore be difficult and lead to multiple, and sometimes invasive tests, such as muscle biopsy. This study aims to describe the diagnoses associated with persistent elevation of serum creatine kinase and to precise the role of the muscule biopsy.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalised in a ward of internal medicin
* having a persistent elevation of serum creatine kinase >3 times the upper normal laboratory value, repeated for 2 times

Exclusion Criteria:

* known neuro-muscular disease causing elevation of creatine kinase
* evident post-traumatic cause responsible for the elevation of creatine kinase
* incomplete medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in the ward of internal medicin of Nancy University Hospital or UNEOS General Hospital of Metz between 2009 and 2018.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Diagnosis | at the end of all investigations, an average of 12 months
  The final diagnosis, as written in the medical record at the end of the investigations in the ward of internal medicin, responsible for the elevation of creatine kinase between: inflammatory myositis, mitochondrial myopathy, muscular dystrophy, non neuromuscular pathology

SECONDARY OUTCOMES:
Muscle biopsy | at the end of all investigations, an average of 12 months
  Among the patients who underwent a muscle biopsy, number of anormal biopsies that contributed to make the final diagnosis responsible of the elevation of creatine kinase
Clinical presentation | at the end of all investigations, an average of 12 months
  association between the initial clinical presentation and the final diagnosis
Paraclinical presentation | at the end of all investigations, an average of 12 months
  association between the initial paraclinical presentation and the final diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France